CLINICAL TRIAL: NCT01090466
Title: A Phase I/II Single-Arm Trial to Evaluate the Combination of Cisplatin and Gemcitabine With the mTOR Inhibitor Temsirolimus for First-Line Treatment of Patients With Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: Gemcitabine Hydrochloride, Cisplatin, and Temsirolimus as First-Line Therapy in Treating Patients With Locally Advanced and/or Metastatic Transitional Cell Cancer of the Urothelium
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000667766; WCTU-TOTEM; ISRCTN31546330; EUDRACT-2007-007615-82; EU-21014; WCTU-SPON-417-07; CRUK-08/015
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: transitional cell carcinoma of the bladder; recurrent bladder cancer; recurrent urethral cancer; recurrent transitional cell cancer of the renal pelvis and ureter; stage IV bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; distal urethral cancer; proximal urethral cancer; urethral cancer associated with invasive bladder cancer; stage IV urethral cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Cisplatin; Gemcitabine; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: temsirolimus
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine hydrochloride and cisplatin together with temsirolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of temsirolimus given together with gemcitabine hydrochloride and cisplatin as first-line therapy in treating patients with locally advanced and/or metastatic transitional cell cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine a safety profile of temsirolimus in combination with cisplatin and gemcitabine hydrochloride, including dose-limiting toxicities (DLTs) and maximum-tolerated dose (MTD) in patients with locally advanced and/or metastatic transitional cell carcinoma of the urothelium. (phase I)
* To determine the recommended dose for the Phase II stage of the trial and subsequent studies. (phase I)
* To assess progression-free survival (PFS) at six months from date of enrollment. (phase II)

Secondary

* To determine the pharmacokinetic profile of temsirolimus in combination with cisplatin and gemcitabine hydrochloride. (phase I)
* To determine tolerability (side-effects) and feasibility (number of participants requiring dose delays or reduction and/or treatment withdrawal). (phase II)
* To determine objective response rate as assessed by RECIST. (phase II)
* To assess PFS of these patients. (phase II)
* To assess overall survival of these patients. (phase II)
* To determine toxicity during and after treatment in these patients. (phase II)

OUTLINE: This is a multicenter, phase I dose-escalation study of temsirolimus followed by a phase II study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, cisplatin IV over 3-4 hours on day 1, and temsirolimus IV over 30 minutes on days 1 or 2, 8 or 9, and 15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Blood specimens may be collected periodically for pharmacokinetic studies.

After completion of study treatment, patients are followed at 6 months and 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the urothelium

  * Pure or mixed histology
  * Upper or lower urinary tract
* Radiologically evaluable* locally advanced and/or metastatic disease not amenable to curative treatment with surgery or radiotherapy, meeting any 1 of the following criteria:

  * T4b, any N, any M
  * Any T, N2-3, any M
  * Any T, any N, M1
* NOTE: *Patients enrolled in the phase II portion of the trial must have radiologically measurable disease.
* No transitional cell cancer for which subsequent radical treatment is being considered with a view to possibly cure the disease
* No history of CNS metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and ALP ≤ 2.5 times ULN
* PT or INR ≤ 1.5
* GFR ≥ 60 mL/min (uncorrected for surface area and measured by isotopic means)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Fit to receive cisplatin-containing combination chemotherapy
* No previous malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or incidental localized prostate cancer
* No known HIV positivity or chronic hepatitis B or C infection
* No symptomatic coronary artery disease, myocardial infarction within the past 6 months, congestive cardiac failure (NYHA class III or IV disease), or uncontrolled or symptomatic cardiac arrhythmia
* No clinically significant bacterial or fungal infection

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior radiotherapy or radiotherapy involving more than 30% of total bone marrow volume
* At least 1 month since prior investigational drug
* No prior systemic therapy for locally advanced or metastatic disease

  * Patients who have received prior neoadjuvant or adjuvant chemotherapy for urothelial cancer (up to 4 courses), completed at least 6 months prior to first documented disease progression are eligible
* No concurrent anticoagulant therapy with warfarin or unfractionated heparin

  * Patients requiring anticoagulation may be entered on study after successful conversion to low molecular weight heparin
* No concurrent medications which have known adverse interactions with the treatment used on this trial (e.g., CYP3A4 inhibitors or inducers in phase I of this trial)
* No prior or concurrent live vaccines (e.g., measles, mumps, rubella, oral polio, Bacille Calmette-Guérin [BCG], yellow fever, varicella, and TY21a typhoid vaccines)
* No concurrent grapefruit juice

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Safety (recommended phase II dose and dose-limiting toxicities) (phase I)
Progression-free survival at 6 months (phase I)

SECONDARY OUTCOMES:
Pharmacokinetics (phase I)
Safety, including tolerability and feasibility (phase II)
Overall survival (phase II)
Progression-free survival (time-to-event) (phase II)
Objective (radiological) response rate according to RECIST criteria (phase II)
Toxicity during and after treatment according to NCI CTCAE v 3.0 (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: John Chester, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom